CLINICAL TRIAL: NCT05649189
Title: A Study of the Differences in Telomere Length Between Patients With and Without Food Addiction
Brief Title: Differences in Length of Telomere in Food Addicted vs Non Food Addicted Persons
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Collaborators: University of Washington (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 0122-21-EP
Record Dates: First submitted 2022-12-03; First posted 2022-12-13 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Food Addiction
MeSH Terms: conditions — Food Addiction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants testing positive for Food Addiction (FA): these participants have tested positive for Food Addiction (FA) at a severe level using the YaleFAS-2 Food Addiction Scale.
  Interventions: Diagnostic Test: telomere length measure
- Participants testing negative for Food Addiction (FA): these participants have tested negative for Addiction (FA) using the YaleFAS-2 Food Addiction Scale.
  Interventions: Diagnostic Test: telomere length measure

INTERVENTIONS:
Diagnostic Test: telomere length measure — length of telomere between two groups

SUMMARY:
The purpose of this descriptive study is to examine telomere length between two groups of people, those with and those without food addiction and identify possible relationships that may play a role in food addiction, it's behaviors and consequences. Research subjects would be adults age 19-70. They would be recruited from the Rural Nebraska Panhandle population. All COVID precautions will be enforced. Human subjects safety plans will be in place for this study.Eligibility: YaleFAS-2 Food Addiction Scale will be used to screen for presence or absence of food addiction. AT a later time, Eligible persons will be given the research consent form to read through and determine if they want to become a participant. If so, they will be consented. The participants will then be assigned an identification number to maintain confidentiality. Intervention: Participants will be given a Oragene saliva DNA collection kit to use and return to investigators. Evaluation:The Oragene saliva DNA collection kit will then be sent in for telomere length testing. Telomere Results will be correlated with food addiction diagnoses and behaviors to identify potential relationships. Follow up: Publication of results

DETAILED DESCRIPTION:
Food Addiction is often accompanied by overweight/obesity and a host of co-morbidities. From previous pilot studies, we have determined it is difficult to treat and behavioral interventions have limited effectiveness. To better understand possible genetic relationships with food addiction, a handful of researchers have begun to examine this proposed relationship. A meta-analysis (Darrow et al., 2016) that reviewed the studies examining the association between psychiatric disorders and telomere length involved 14,827 persons. Additionally, Daubenmier et al. (2012) examined the relationships among stress, eating, and metabolic factors with telomerase activity with 47 overweight/obese women. These studies lead us to seek proof of concept, that there may be a relationship between food addiction and telomere length and to better characterize persons with and without Food Addiction to enable us to develop interventions specific to each group. In this pilot we will attempt to provide additional scientific knowledge to confirm/support or negate the hypothesis that telomere length may be related to/contributing to Food Addiction. Davis (2019) conducted a review of literature involving food addiction and genetics. In the review, it is noted that thus far there has been only one study that has assessed whether genetic determinants of food addiction overlapped with drug addiction. Two loci (rs75038630 and 74902201) met GW-significance. However, neither of those loci has previously been associated with eating behaviors. We will examine telomere length in our pilot to provide additional evidence for this gap in the knowledge.

The liquid saliva sample kit that will be used is the Oragene saliva DNA collection kit. See following for more specific information.A 2 mL sample of liquid saliva will be obtained by participants spitting into the Oragene saliva DNA collection kit (Genotek Inc. Ottawa, ON, Canada) containing 1 mL of DNA stabilizing liquid. The samples will stored at room temperature until processing for DNA extraction. The saliva samples will be shipped to a laboratory at the University of California San Francisco where the telomere length will be measured by using the monoplex quantitative polymerase chain reaction (qPCR) method. This method has been validated against the Southern blot method. Stout et al. (2017) ran the inter-assay variability test and found that the average coefficient of variation was 2.7% for saliva DNA. Both the saliva collection kit and the telomere length measurement are used only for research purposes (i.e., not commercially available). Stout et al. (2017) report that salivary telomere length was correlated with whole blood telomere length (r = 0.56, p = 0.005).

ELIGIBILITY:
Inclusion Criteria:

* Obese Food addicted persons between ages 19 and 70
* Obese Non Food addicted persons between ages 19 and 70

Exclusion Criteria:

* persons with active liver disease
* persons with active cancer

Ages: 19 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All those enrolled (n = 120) were adults (age 19-70) with overweight/obesity (BMI ≥ 25). Half were positive for severe FA (≥ 6 symptoms plus clinical significance) and half were negative for FA (≤ 1 symptom and no clinical significance). These criteria were selected to best define the FA+ and FA- subtypes (Aguirre et al., 2022). Most participants were female (87.5%) and Caucasian (65%). The remainder were Latino (24%), African American (7%), Asian (4%), or Native American (2%). Reported health conditions include diabetes (n = 5), hypertension (n = 20), smoking (n = 4).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-10-17 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
telomere length | at baseline only
  cross sectional saliva sample from which telomere length is measured

CONTACTS AND LOCATIONS:
Overall Officials: Trina M Aguirre, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, College of Nursing, Scottsbluff, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
Group data will be shared via publication.Genetic data will not be shared with individuals or other researchers.